CLINICAL TRIAL: NCT05275530
Title: The Impact of Choice on Colorectal Cancer (CRC) Screening Uptake Among Average-risk Individuals 45-49 Years of Age
Brief Title: The Impact of Choice on Colorectal Cancer Screening
Acronym: CRC45+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: UCLA Vatche and Tamar Manoukian Division of Digestive Diseases (Unknown)
Responsible Party: Principal Investigator, Daniel M. Croymans, MD, MBA, MS, Medical Director, DOM Quality, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRC45
Record Dates: First submitted 2022-02-19; First posted 2022-03-11 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Health Screening
Keywords: Colorectal Cancer Screening; Choice
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: * Parallel-arm randomized controlled trial
  * Patient-level randomization
  * Four arms
    * Arm 0: Standard of care control
    * Arm 1: Active FIT choice
    * Arm 2: Active colonoscopy choice
    * Arm 3: Active FIT v. colonoscopy choice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (No Intervention): No Intervention-"Standard Care"
  UCLA Health has a mailed FIT outreach program. This group will receive standard FIT mailer protocol. They will receive a tailored MyChart message indicating the importance of CRC screening and not be presented with a choice for screening modalities.
- FIT Choice (Experimental): This group will receive a tailored message via MyChart with information about CRC screening and using the FIT kit for noninvasive screening. They will then have to actively choose if they want CRC screening with a FIT kit vs no screening. If they opt for screening, the investigators will mail them a FIT kit.
  Interventions: Behavioral: Active FIT Choice
- Colonoscopy Choice (Experimental): This group will receive a tailored message via MyChart with information about CRC screening and colonoscopy for CRC screening. They will then have to actively choose if they want CRC screening with a colonoscopy vs no screening. If they opt for screening, the investigators will direct them to our patient navigators to get scheduled for a colonoscopy.
  Interventions: Behavioral: Active Colonoscopy Choice
- Dual Choice (Experimental): This group will receive a tailored message via MyChart with information about CRC screening and using either the FIT kit or colonoscopy for CRC screening. They will then have to actively choose if they want CRC screening with a FIT kit, a colonoscopy, or no screening. If they opt for screening, the investigators will either mail them a FIT kit or direct them to our patient navigators to schedule a colonoscopy, depending on their choice.
  Interventions: Behavioral: Active Dual Choice

INTERVENTIONS:
Behavioral: Active FIT Choice — The investigators will send randomized participants a message via MyChart indicating the benefits of CRC screening, along with tailored information about FIT as a screening strategy. At the end of the message, participants will complete a survey asking them to indicate if they would like to be screened for CRC with a FIT, or if they prefer no screening whatsoever. The investigators will then ask follow-up questions to better understand the reason patients made their respective choices.
  Arms: FIT Choice
Behavioral: Active Colonoscopy Choice — The investigators will send randomized participants a message via MyChart indicating the benefits of CRC screening, along with tailored information about colonoscopy as a screening strategy. At the end of the message, participants will complete a survey asking them to indicate if they would like to be screened for CRC with a colonoscopy, or if they prefer no screening whatsoever. The investigators will then ask follow-up questions to better understand the reason patients made their respective choices.
  Arms: Colonoscopy Choice
Behavioral: Active Dual Choice — The investigators will send randomized participants a message via MyChart indicating the benefits of CRC screening, along with tailored information about FIT Kit and Colonoscopy screening. At the end of the message, participants will complete a survey asking them to indicate if they would like to be screened for CRC with either a FIT or Colonoscopy, or if they prefer no screening whatsoever. The investigators will then ask follow-up questions to better understand the reason patients made their respective choices.
  Arms: Dual Choice

SUMMARY:
In May of 2021, the United States Preventive Service Task Force (USPSTF) updated their colorectal cancer (CRC) screening guidelines by recommending screening at an earlier age for average-risk adults starting at the age of 45 years old (Grade B recommendation). This is in addition to their Grade A recommendations of continuing to screen average-risk adults ages 50-75 years old. UCLA Health previously implemented a fecal immunochemical test (FIT) outreach program wherein FIT kits are mailed to average-risk patients overdue for CRC screening twice annually to promote screening uptake. As the investigators health system aims to screen the newly eligible population of average-risk patients between the ages of 45-49, the investigators proposed randomized controlled trial is aimed to determine the most effective patient outreach approach to maximize screening uptake within this age-group.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer-related death for both men and women in the United States. One in 17 Americans will suffer from CRC during their lifetime and early detection of cancers and polyps by screening is shown to reduce CRC mortality. In 2021, the USPSTF updated its CRC screening guidelines to start screening average-risk individuals at the age of 45 years due in part to a rising incidence of CRC and premalignant polyps in younger patients.

Conventional screening options include both invasive (or direct-visualization) and non-invasive (or stool-based) options. Invasive screening tests include flexible sigmoidoscopy, CT colonography, and colonoscopy. Non-invasive screening tests include the fecal immunochemical test (FIT), the high sensitivity guaiac fecal occult blood test, and stool DNA testing. All of these screening tests are recommended by the USPSTF for CRC screening.

Nationally (and at UCLA Health), the two most common CRC screening modalities are the colonoscopy and the FIT. UCLA Health has previously implemented a FIT mailer outreach program wherein FIT kits are mailed to average-risk patients overdue for CRC screening twice annually to promote screening uptake. The program has been extremely effective in increasing CRC screening adherence rates, with an increase in the health system's screening rate over the past several years.

The investigators current study aims to determine the most effective patient outreach approach to maximize CRC screening utilization in average-risk individuals ages 45-49 years. In addition, the investigators aim to understand the impact of screening modality choice on uptake of CRC screening, patients' preference for screening modality, and sociodemographic differences in screening utilization among individuals ages 45-49 years.

There are approximately 18,000 patients eligible for inclusion. The investigators will randomly assign approximately 17,000 average-risk patients aged 45-49 to one of four arms. 1,000 of the patients will be reserved for an internal pilot project. In all arms, all patients will receive a text message encouraging them to access their patient communication portal via Epic electronic health record (EHR) (referred to as "MyChart"). In all arms, once a patient visits MyChart, a message on MyChart will state that they are due for CRC screening and the importance of CRC screening. In the control (standard care) arm, patients will treated as part of our "FIT-kit mailer program." These patients will receive a mailed FIT kit, and the message on MyChart will encourage them to complete the FIT kit. In the "FIT Kit Choice" arm, patients will be presented with the choice to complete screening with a FIT kit or opt out of screening. In the "Colonoscopy Choice" arm, patients will be presented with the choice to complete screening with a colonoscopy or opt out of screening. In the "Dual Choice" arm, patients will be presented with the choice to complete screening with a FIT kit, complete screening with a colonoscopy, or opt out of screening. After patients make the choice in MyChart, the patient will be asked why they made that choice.

We will resend the message on MyChart (as a reminder) two weeks after they receive the initial MyChart message. The reminder message content will be very similar to the content of initial MyChart message, and differ by arm.

The investigators have competing predictions based on the literature about whether giving people the option of choosing between two screening modalities (vs. neither) is better than giving people the option of deciding whether to take one modality (vs. not). On the one hand, offering people two modalities should increase flexibility and thus enhance participation; on the other hand, choosing between two modalities could tax mental resources and create choice avoidance, thus decreasing participation. Specifically:

In addition, the investigators have competing predictions based on the literature about whether active choice is better than assigning people a screening modality. On one side, active choice can make patients feel more empowered, thus enhancing participation in screening. On the other side, active choice takes more of patients' cognitive and time resources than following the assigned option, thus decreasing participation in screening.

Analysis Plan:

* Patient-level linear regression models with robust standard errors
* The primary model term will be indicator variables for arms that patients are assigned to.
* Covariates will include age, sex, race/ethnicity, social vulnerability index (ZIP code level), and baseline HM focus measure completion rate
* Treatment effects will be summarized using rate differences and 95% confidence intervals
* Exploratory analyses will investigate heterogeneous treatment effects by splitting the sample into demographic subgroups and by testing for demographic x choice arm interactions
* Sensitivity analyses will be performed without covariates, and using logistic regression models in place of linear regression models
* Missing covariate values will be handled by including 'unknown' indicators, along with mean imputation for quantitative covariates
* To analyze the effect of offering a choice between modalities (vs. single choice), we will compare the single choice arms (arms 1 and 2) with the dual choice arm (arm 3).
* To analyze the effect of active choice, we will compare the control arm (arm 0) with (1) active FIT choice arm (arm 1) and (2) the dual choice arm (arm 3).
* To assess both the effect of offering the dual choice (vs. single choice) and the effect of active choice, we will analyze two samples: (1) patients who open their initial MyChart message within 1 week of the date sent and (2) intention-to-treat regardless of whether patients open the MyChart message. In addition, when assessing the effect of offering the dual choice (vs. single choice), we will also examine patients who open either the initial or the reminder MyChart message within 1 week.

ELIGIBILITY:
Inclusion Criteria

* UCLA Health patient
* Age 45-49 (as of 1/1/2022)
* Active primary care provider at UCLA Health
* Visit within the last 3 years

Exclusion Criteria

* Age <45 or >50 years old at time of randomization
* Documented family history of CRC in EMR
* History (personal or family) of prior adenomatous polyps in the EHR
* History of high-risk cancer syndromes (e.g., Lynch, FAP)
* Prior CRC screening with colonoscopy or FIT
* Inactive MyChart status at enrollment
* No documented SMS-capable phone number

Ages: 45 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20509 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Overall completion of any Colorectal Cancer Screening test | 6 months after getting the text message
  Rate of completion of any CRC screening (FIT Kit or Colonoscopy) throughout the observation window.

SECONDARY OUTCOMES:
Selection of modality in MyChart Survey | within 4 weeks from receiving the initial MyChart message
  Frequency of CRC screening choice indicated in the MyChart survey per arm
CRC screening order placed by any modality | within 6 weeks from receiving the initial MyChart message
  The frequency of ordering FIT Kit or Colonoscopy in the "FIT Kit Choice", "Colonoscopy Choice" and "Dual Choice" arms
Colorectal cancer screening uptake by modality | 6 months after getting the initial MyChart message
  Rate of completion of CRC screening by specific modality (FIT Kit or Colonoscopy) throughout the observation window.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Health Department of Medicine, Quality Office, Los Angeles, California
  - UCLA Vatche and Tamar Manoukian Division of Digestive Diseases, Westwood, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No
We do not plan to make any individual participant data available.

REFERENCES:
- [Derived] Galoosian A, Dai H, Croymans D, Saccardo S, Fox CR, Goshgarian G, De Silva S, Han MA, Vangala S, May FP. Population Health Colorectal Cancer Screening Strategies in Adults Aged 45 to 49 Years: A Randomized Clinical Trial. JAMA. 2025 Sep 2;334(9):778-787. doi: 10.1001/jama.2025.12049. PMID 40758331